CLINICAL TRIAL: NCT06887933
Title: A Prospective, Multicentre, Open Labelled, Single Arm Phase-IV Clinical Trial of Niraparib in Indian Patients With Advanced or Relapsed Ovarian Cancer Who Are in Complete or Partial Response Following Platinum Based Chemotherapy
Brief Title: A Trial to Evaluate the Safety of Niraparib Tablets in Adult Female Participants With Advanced or Relapsed Epithelial Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 220168
Record Dates: First submitted 2025-03-19; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Neoplasms
Keywords: Niraparib; Ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Niraparib (Experimental)
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib will be administered.

SUMMARY:
The goal of this clinical trial is to learn about the safety profile of niraparib in adult female participants for the treatment of advanced or relapsed epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female participants with ≥18 years of age, able to understand the study procedures and agree to participate in the study by providing written informed consent.
* Histologically confirmed epithelial ovarian cancer.

  * Eligible for active study drug treatment according to the approved label - as monotherapy for the maintenance treatment of adult participants with advanced epithelial (International Federation of Gynecology and Obstetrics [FIGO] stage III and IV) high-grade ovarian, fallopian tube or primary peritoneal cancer who are in response (complete or partial) following completion of first-line platinum-based chemotherapy.
  * as monotherapy for the maintenance treatment of adult participants with platinum-sensitive relapsed high grade serious epithelial ovarian, fallopian tube, or primary peritoneal cancer who are in response (complete or partial) to platinum-based chemotherapy.
* Laboratory complete blood count (CBC) criteria (Absolute neutrophil count ≥1,500/microliters [μL]; Platelets ≥100,000/μL; Hemoglobin ≥9 grams per decilitre [g/dL]).
* Adequately controlled hypertension basis on investigator's discretion.
* Women of childbearing potential must be ready to use contraceptive measures to avoid pregnancy during study period and until 180 days after the last dose.

Exclusion Criteria:

* Participant is pregnant, breastfeeding, or expecting to conceive children while receiving study treatment and for up to 180 days after the last dose of study treatment.
* Participant had known, active hepatic disease, known case of end-stage renal disease (ESRD), known case of serious, uncontrolled medical disorder, any known history or current diagnosis of Myelodysplastic syndrome (MDS) or Acute myeloid leukemia (AML).
* Any previous polymerases inhibitor (PARPi) treatment.
* Participant with concomitant serious uncontrolled medical illness.
* Participant is receiving niraparib for use that is not according to the approved label.
* Participant with either the history of hypersensitivity to excipients of the study drug or to drugs with a similar chemical structure or class to the study drug.
* Participant with a previously or currently diagnosed MDS/ AML or pneumonitis.
* Participants who have not recovered sufficiently from prior surgery or anticancer treatment.
* Participants who have known history of hepatitis B or hepatitis C.
* Participant with active infection such as tuberculosis (TB) Prior/concurrent clinical study experience.
* Participation in another clinical study with a study drug administered in the last 3 months.
* Judgment by the investigator that the participant should not take part in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.
* Previous enrolment in the present study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 67 (Estimated)
Dates: Start 2025-04-22 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-07-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to Day 105

SECONDARY OUTCOMES:
Number of participants with serious adverse events (SAEs), TEAEs leading to death, TEAEs leading to dose reduction, TEAEs leading to treatment discontinuation | Up to Day 105

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/